CLINICAL TRIAL: NCT03948854
Title: Implementing a Low FODMAP Diet in Irritable Bowel Syndrome Patients: Which Educational Method Works Best
Brief Title: Implementing a Low FODMAP Diet in Irritable Bowel Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian E. Lacy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-011391
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Registered dietitian education (Experimental): Subjects with irritable bowel syndrome (IBS) will receive education on FODMAP diet in person by a registered dietitian
  Interventions: Other: Registered dietitian
- On-line video program education (Experimental): Subjects with irritable bowel syndrome (IBS) will receive education on FODMAP diet using an on-line video program
  Interventions: Other: On-line video program
- Handout education (Experimental): Subjects with irritable bowel syndrome (IBS) will receive education on FODMAP diet by a printed handout
  Interventions: Other: Printed handout
- Dietitian-led group education (Experimental): Subjects with irritable bowel syndrome (IBS) will receive education on FODMAP diet in a dietitian-led group setting
  Interventions: Other: Dietitian-led group

INTERVENTIONS:
Other: Registered dietitian — Education on low FODMAP diet is provided in person by a registered dietitian who is an expert on the low FODMAP diet
  Arms: Registered dietitian education
Other: On-line video program — Education on low FODMAP diet is provided by an on-line program via a link sent through email
  Arms: On-line video program education
Other: Printed handout — Education on low FODMAP diet is provided through printed handout material at the initial visit.
  Arms: Handout education
Other: Dietitian-led group — Education on low FODMAP diet is provided in a dietitian-led group setting
  Arms: Dietitian-led group education

SUMMARY:
Researchers are trying to determine the best course of action regarding the dietary management with a diet low in fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP diet) for irritable bowel syndrome.

DETAILED DESCRIPTION:
An analysis of different educational programs providing information on the low FODMAP diet will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-75 years) seen in the primary care clinic or in the Gastroenterology clinic at Mayo Clinic Florida, who are diagnosed with IBS by Rome IV criteria

Exclusion Criteria:

* Subjects who have previously tried the low FODMAP diet (whether successful or not)
* Current or recent (less than 4 weeks) opioid use
* Current or recent (less than 10 weeks) rifaximin use
* Inability to speak or read English
* Pregnancy and/or breast-feeding
* Medical or psychological issues that would prevent modifying their diet for 8 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Improvement in IBS symptoms | Baseline, end of study approximately 8 to 10 weeks
  Change in IBS symptoms will be measured from baseline to the end of study using the validated IBS symptoms severity scale (IBS-SS). This is a visual analog scale from 0-100. The primary outcome measure is improvement in symptom scores from end of study to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lacy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials